CLINICAL TRIAL: NCT05230355
Title: Comparison Between Two Techniques of Subthreshold Diode Laser Cyclophotocoagulation in Refractory Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Omar, Assistant lecturer of ophthalmology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTTSDLCRG
Record Dates: First submitted 2022-01-20; First posted 2022-02-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2022-01

CONDITIONS: Refractory Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A the standard technique (Active Comparator): The tip of the probe was moved in a "painting" motion along the upper and lower hemispheres over pars plana, 3 mm behind the limbus, avoiding the 3 and 9 o'clock positions.
  Interventions: Device: standard technique
- Group B a modified technique (Active Comparator): The probe tip was moved for 2 mm perpendicular to a line 3 mm parallel to the cornea, aiming to cover the largest circumference of the ciliary body area.
  Interventions: Device: modified pattern

INTERVENTIONS:
Device: standard technique — The probe was moved over each hemisphere for 120 seconds (a total of 240 seconds). Total energy = 2.5 x 0.313 x 240 = 187.8 J
  Arms: group A the standard technique
Device: modified pattern — The probe was moved over 3 quadrants for 80 seconds for each quadrant (a total of 240 seconds). Total energy = 2.5 x 0.313 x 240 = 187.8 J
  Arms: Group B a modified technique

SUMMARY:
The aim of this study is to assess the results of subliminal subthreshold transscleral diode cyclophotocoagulation in refractory glaucoma using the standard technique of 360 degree application and to compare the outcome with a modified technique both in terms of efficacy and safety.

DETAILED DESCRIPTION:
Refractory glaucoma is glaucoma that doesn't respond favorably to surgical and/or medical treatment to lower intraocular pressure. It can include primary open angle glaucoma, primary angle closure glaucoma, neovascular glaucoma or silicone oil-induced glaucoma. Cyclophotocoagulation (CPC) is a form of cycloablation using laser to treat glaucoma. It involves ciliary body destruction by targeting the ciliary epithelium and stroma, resulting in a reduction in aqueous secretion and hence intraocular pressure. Transscleral cyclophotocoagulation using a continuous diode laser has been a treatment option in advanced glaucoma cases with s¬¬uboptimal IOP control, for a long time. High treatment energy used by diode laser cyclophotocoagulation was argued to be associated with increased frequency of serious complications such as vision loss, hypotony, and phthisis. These concerns necessitate modulation of the parameters of laser treatment used.

Micropulse transscleral cyclophotocoagulation (MP-TSCPC), which is a variation of conventional continuous-wave CPC, has emerged as an attractive alternative for the treatment of many types of glaucoma. It breaks the continuous wave laser into multiple short and repetitive pulses that allow the tissue to cool down between applications, thus reducing thermal damage. This strategy delivers very short energy pulses followed by rest periods, which is known as "duty cycle" and is defined as the ratio of time that a laser is delivering energy vs resting (ON/OFF). For this procedure, an infrared diode laser is used to stimulate the ciliary body structures and the uveoscleral pathway. This way it reduces the production of the aqueous humour and facilitates the uveoscleral outflow, with IOP reduction as a final effect.

Despite promising results, only few clinical studies are published on MP-TSCPC and most of them are retrospective studies refer to patients having previous continuous wave transscleral cyclophotocoagulation. Moreover, Several parameters and protocols have been studied in other reports in an attempt to refine the standard technique aiming to improve the outcomes without increasing the adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* patients with refractory glaucoma (IOP > 21 mmHg unresponsive to maximally tolerated antiglaucoma medications, previously failed surgical treatment, or both)

Exclusion Criteria:

* Ocular inflammation.
* Ocular infection.
* Recent ocular surgery in the study eye in the 2 months prior to enrolment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
IOP reduction success rate | 6 months
  Success rate is defined as achieving an IOP between 5 and 21 mmHg or at least a 20% reduction in IOP at the final follow up with or without IOP lowering medications

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No